CLINICAL TRIAL: NCT03387553
Title: A Pilot Study Utilizing a HER2 Directed Dendritic Cell Vaccine During Neoadjuvant Therapy of HER2+ Breast Cancer
Brief Title: HER2 Directed Dendritic Cell Vaccine During Neoadjuvant Therapy of HER2+Breast Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19337
Record Dates: First submitted 2017-12-19; First posted 2018-01-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Cancer, Male; Invasive Breast Cancer; HER2-positive Breast Cancer; HER2 Positive Breast Carcinoma; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Immunotherapy; Dendritic Cell Vaccine; DC1
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Immunotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: The trial will consist of two phases. The first lead in phase will enroll 12 participants evenly divided into two arms (alternating enrollment) with different initial priming vaccination schedules.
  Following accrual of this initial group of 12 patients, HER2 ELISPOT post vaccination responses will be assessed to determine which of the two sequences provides the greater increase in anti HER2 response at week 4 over baseline. This will determine which sequence will be used in the second expansion phase of accrual. If both arms are determined equal then Arm A will be selected as the default sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead In Phase - Arm A (Active Comparator): Arm A: One Dendritic Cell Vaccine (DC1) per week x 3 weeks.
  Interventions: Biological: Dendritic Cell Vaccine (DC1); Drug: Neoadjuvant Chemotherapy; Procedure: Curative Surgery
- Lead In Phase - Arm B (Active Comparator): Arm B: Two DC1 vaccinations per week (given 3 days apart i.e., Mon and Thurs or Tues and Friday) x 3 weeks.
  Interventions: Biological: Dendritic Cell Vaccine (DC1); Drug: Neoadjuvant Chemotherapy; Procedure: Curative Surgery
- Expansion Phase (Experimental): DC1 vaccinations according to optimal vaccination schedule. Participants will receive a booster intranodal study vaccine at week 25 prior to receiving surgery. Participants will then undergo definitive curative surgery following completion of the neoadjuvant therapy, additional adjuvant locoregional/systemic therapy (as deemed appropriate by their treating physicians).
  Interventions: Biological: Dendritic Cell Vaccine (DC1); Drug: Neoadjuvant Chemotherapy; Procedure: Curative Surgery

INTERVENTIONS:
Biological: Dendritic Cell Vaccine (DC1) — Study Vaccine:
  Lead In Phase - Weekly as outlined in each treatment Arm.
  Expansion Phase - At the optimal schedule determined at the end of the Lead In Phase.
  Pre-surgery - Booster Vaccine at week 25 prior to receiving surgery.
  Post-surgery - Participants will receive a series of 3 booster intranodal study vaccines given once every 6 months.
  Other Names: Immunotherapy
Drug: Neoadjuvant Chemotherapy — Upon completion of the 3 week series of vaccinations participants will then undergo neoadjuvant chemotherapy treatment with the TCH-P Taxotere (docetaxel), Carboplatin, Herceptin (trastuzumab), Perjeta (pertuzumab) standard of care neoadjuvant chemotherapy regimen given intravenously once every 3 weeks for up to 6 cycles. The treating physician will have the discretion to delay, modify, or shorten the neoadjuvant chemotherapy as per routine practice guidelines and physician discretion.
  Other Names: TCHP
Procedure: Curative Surgery — Planned definitive curative surgery at 26 to 28 weeks.

SUMMARY:
The purpose of this study is to learn more about how to treat patients with HER-2/neu positive invasive breast cancer (IBC). HER-2/neu is a type of protein that is known to be over-expressed in aggressive breast cancer.

The study drug for this trial is DC1 study vaccine which is a HER2-sensitized dendritic cell (DC) study vaccine. This study vaccine is made from the participant's blood cells collected from a procedure called leukapheresis. Dendritic cells are immune cells that can tell the immune system to fight infection. In laboratory testing and from previous studies in participants, these cells may also help the immune system attack tumors such as breast cancer.

DETAILED DESCRIPTION:
The trial will consist of two phases. The first lead in phase will enroll 12 participants evenly divided into two arms (alternating enrollment) with different initial priming study vaccination schedules.

Arm A: One DC1 study vaccination per week x 3 weeks. Arm B: Two DC1 study vaccinations per week (given 3 days apart for example Mon and Thurs or Tues and Friday) x 3 weeks.

Following accrual of this initial group of 12 participants, HER2 ELISPOT post study vaccination responses will be assessed to determine which of the two sequences provides the greater increase in anti HER2 response at week 4 over baseline. This will determine which sequence will be used in the second expansion phase of accrual. If both arms are determined equal then Arm A will be selected as the default sequence.

Second phase of accrual will consist of 14 additional participants to undergo study vaccination using the optimal schedule declared in the first phase of the trial. The trial will consist of two phases. The first lead in phase will enroll 12 participants evenly divided into two arms (alternating enrollment) with different initial priming study vaccination schedules.

Arm A: One DC1 study vaccination per week x 3 weeks Arm B: Two DC1 study vaccinations per week (given 3 days apart for example Mon and Thurs or Tues and Friday) x 3 weeks.

Following accrual of this initial group of 12 participants, HER2 ELISPOT post study vaccination responses will be assessed to determine which of the two sequences provides the greater increase in anti HER2 response at week 4 over baseline. This will determine which sequence will be used in the second expansion phase of accrual. If both arms are determined equal then Arm A will be selected as the default sequence.

Second phase of accrual will consist of 14 additional participants to undergo study vaccination using the optimal schedule declared in the first phase of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed clinical stage II or III ERPR- HER2+ (per CAP criteria) invasive carcinoma of the breast
* Medically and surgically appropriate to undergo neoadjuvant chemotherapy with TCH-P Taxotere (docetaxel), Carboplatin, Herceptin (trastuzumab), Perjeta (pertuzumab) regimen followed by standard of care local therapy as determined by their treating physician
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than 2
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits - OR -
  * creatinine clearance ≥60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction within institutional normal limits by either MUGA or ECHO at baseline.
* Women of child-bearing potential and their male partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Sexually active male participants should use a barrier method or exercise abstinence during chemotherapy administration until surgery.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with inflammatory breast cancer, widespread locally advanced unresectable disease involving the chest wall/nodal basins in which a curative surgical resection cannot be performed, or those in whom de novo metastatic disease is suspected or confirmed
* May not be receiving any other investigational agents for the treatment of their breast cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study vaccine components and any of the chemotherapy drugs (docetaxel, carboplatin, trastuzumab, pertuzumab)
* Unwilling or unable to undergo an apheresis for production of their vaccine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breastfeeding
* Known congenital or acquired immune deficiency (including those patients who require systemic immunosuppressant drugs for autoimmune disease or organ transplant).
* Pre-existing peripheral neuropathy that would limit treatment with taxanes and platinum agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Expansion Phase Schedule Selection by Week 4 | By Week 4
  Immunogenicity of HER2 DC Vaccine per treatment Arm, based on week 4 ELISPOTs. Three metrics of CD4+ Th1 response will be computed for each patient, (a) overall anti-HER2 responsivity (i.e., if patient demonstrates a positive ELISPOT response to >1 peptide, (b) response repertoire (i.e., number of reactive peptides) and (c) cumulative response (total SFC/10^6 cells across 6 peptides). The primary immunogenicity outcome will be the cumulative response at week 4 (week after completion of all vaccinations).
Pathologic Complete Response (pCR) Rate | Week 26 to 28 - At post-surgical pathological assessment
  Pathologic complete response rate of participants treated in the Expansion Phase. Clinical efficacy will be defined by the pathologic complete response (pCR) rate, the percentage of patients who achieve pCR based on surgical pathology assessment.The definition of pathologic complete response (pCR) will be ypT0/is N0 (no residual viable invasive disease in the breast or nodes). Any response less than pCR will be scored as incomplete response or progression (if tumor size increases during neoadjuvant chemotherapy on physical exam/breast imaging).

SECONDARY OUTCOMES:
Recurrence Free Survival (RFS) | Up to 3 years post-surgery
  Recurrence-free survival (RFS) will be defined as the time from first vaccination to documented recurrence (any breast event), death due to any cause or last patient contact that documents recurrence-free status (i.e., a clinic or scan date).

CONTACTS AND LOCATIONS:
Overall Officials: Haten Soliman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Soliman H, Aldrich A, Abdo N, Han H, Soyano A, Costa R, Armaghani A, Kiluk J, Khakpour N, Lee MC, Hoover S, Laronga C, Niell B, Mooney B, Weinfurtner RJ, Rosa M, Czerniecki B. A pilot study incorporating HER2-directed dendritic cells into neoadjuvant therapy of early stage HER2+ER- breast cancer. NPJ Breast Cancer. 2025 Mar 17;11(1):29. doi: 10.1038/s41523-025-00742-x. PMID 40097486
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/